CLINICAL TRIAL: NCT00228579
Title: Assessment of Changes in Abdominal Fat and Metabolic and Tissue Biomarkers During a Bariatric Surgery Weight Loss Intervention Program
Brief Title: Assessment of Changes in Abdominal Fat
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nana Gletsu Miller, Assistant Professor, Foods and Nutrition, Indiana University
Other Study IDs: 333-2002; DK-067167
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Obesity
Keywords: diabetes; insulin resistance
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bariatric Surgery: Subjects will be recruited from patients undergoing bariatric surgery at Emory Bariatrics. The cost of surgical procedures will not be provided by the research study.

SUMMARY:
In this study, we propose to determine the effect of weight loss on amount of body fat, and on body fat distribution, in severely obese patients. We also want to determine what measurements (waist, hip or thigh circumference) best show the changes in body fat and fat distribution in this group. Most importantly, we want to relate the changes in body measurements to changes in health indicators (blood cholesterol, blood pressure, blood sugars, liver function). With the findings of this study, clinicians should be able to predict an improvement in health based on a change in waist, hip or thigh size. Because this is a pilot study, we will focus on women, who make up the bulk of our clinic population. We will also focus on racial differences between Caucasians and Blacks.

DETAILED DESCRIPTION:
Severe obesity affects 4.7% of the U.S. population. A significant number of these individuals suffer from impaired glucose tolerance and type II diabetes due to insulin resistance (IR). Although it is generally accepted that the accumulation of intraabdominal (IA) fat increases the risk of developing IR, the mechanisms responsible for this phenomenon are not yet understood. In addition, the role of subcutaneous (SC) fat towards the etiology of IR - protective, inert or detrimental - is still under debate. This is because SC adipose tissue releases adipocytokines (IL-6, leptin, TNF-a) that have been demonstrated to impair insulin action. In individuals who are severely obese, hyperinsulinemia may induce an exaggerated production of adipocytokines from IA compared to SC fat stores. Our specific aims are: (1) to determine relative contribution of abdominal SC fat versus IA fat to systemic levels of IL-6, leptin and TNF-a in lean and in severely obese individuals; (2) to determine the effects of systemic adipocytokine concentrations on whole body as well as tissue sensitivity to insulin. Hypothesis: (a) In the context of severe obesity, IA fat produces increased quantities of IL-6, leptin and TNF-a compared to SC fat; (b) In severely obese patients undergoing weight loss, whole body and tissue IR can be predicted by changes in systemic adipocytokines. Methods: Adipose tissue content of IL-6, leptin and TNF-a will be determined by ELISA in biopsies obtained from IA and SC fat stores in lean and severely obese patients. Computer tomography-determined areas of IA and SC fat will be related to changes in systemic adipocytokines at baseline and 6-mo following weight loss therapy. Changes in systemic IL-6, leptin and TNF-a will be assessed from measurements made at baseline and following 6-mo weight loss. For this time period we will also determine changes in whole body (via IVGTT) and tissue sensitivity to insulin (via glucose uptake into muscle and fat). Relationships between systemic adipocytokines and IR will be assessed using uni- and multivariate correlation analysis. These novel studies will determine whether hypersecretion of adipocytokines by IA versus SC adipose tissue induces IR in patients with severe obesity.

ELIGIBILITY:
Exclusion Criteria:

1. male [this will be a pilot study limited to females. Gender is known to influence adipose tissue distribution and females represent the majority of the Emory Bariatrics population - 89%],
2. age less than 18 or greater than 65 y, [aging has been independently associated with insulin resistance]
3. pregnancy
4. not eligible for treatment due to medical history (due to cardiac, hepatic or psychiatric problems, or immunocompromise),
5. tobacco smoker

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severely obese volunteers who are undergoing bariatric surgery. Subjects will be recruited from patients who are undergoing bariatric surgery procedures at Emory Bariatrics. The costs of surgical procedures are not provided by the research study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2003-06; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Visceral adipose tissue volume | Baseline, 1, 6 and 24 months
  Visceral adipose tissue volume is measured by computed tomography

SECONDARY OUTCOMES:
Insulin sensitivity | Baseline, 1, 6, 24 months
  Insulin sensitivity is measured by intravenous glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Nana Gletsu Miller, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Background] Gletsu-Miller N, Hansen JM, Jones DP, Go YM, Torres WE, Ziegler TR, Lin E. Loss of total and visceral adipose tissue mass predicts decreases in oxidative stress after weight-loss surgery. Obesity (Silver Spring). 2009 Mar;17(3):439-46. doi: 10.1038/oby.2008.542. Epub 2008 Dec 11. PMID 19219062
- [Result] Lin E, Liang Z, Frediani J, Davis SS Jr, Sweeney JF, Ziegler TR, Phillips LS, Gletsu-Miller N. Improvement in ss-cell function in patients with normal and hyperglycemia following Roux-en-Y gastric bypass surgery. Am J Physiol Endocrinol Metab. 2010 Nov;299(5):E706-12. doi: 10.1152/ajpendo.00405.2010. Epub 2010 Aug 17. PMID 20716694
- [Result] Lin E, Phillips LS, Ziegler TR, Schmotzer B, Wu K, Gu LH, Khaitan L, Lynch SA, Torres WE, Smith CD, Gletsu-Miller N. Increases in adiponectin predict improved liver, but not peripheral, insulin sensitivity in severely obese women during weight loss. Diabetes. 2007 Mar;56(3):735-42. doi: 10.2337/db06-1161. PMID 17327444
- [Result] Gletsu-Miller N, Kahn HS, Gasevic D, Liang Z, Frediani JK, Torres WE, Ziegler TR, Phillips LS, Lin E. Sagittal abdominal diameter and visceral adiposity: correlates of beta-cell function and dysglycemia in severely obese women. Obes Surg. 2013 Jul;23(7):874-81. doi: 10.1007/s11695-013-0874-6. PMID 23408092
- [Result] Gletsu-Miller N, Broderius M, Frediani JK, Zhao VM, Griffith DP, Davis SS Jr, Sweeney JF, Lin E, Prohaska JR, Ziegler TR. Incidence and prevalence of copper deficiency following roux-en-y gastric bypass surgery. Int J Obes (Lond). 2012 Mar;36(3):328-35. doi: 10.1038/ijo.2011.159. Epub 2011 Aug 30. PMID 21876546
- [Result] Lin E, Armstrong-Moore D, Liang Z, Sweeney JF, Torres WE, Ziegler TR, Tangpricha V, Gletsu-Miller N. Contribution of adipose tissue to plasma 25-hydroxyvitamin D concentrations during weight loss following gastric bypass surgery. Obesity (Silver Spring). 2011 Mar;19(3):588-94. doi: 10.1038/oby.2010.239. Epub 2010 Oct 14. PMID 20948527
- [Derived] Forbes R, Gasevic D, Watson EM, Ziegler TR, Lin E, Burgess JR, Gletsu-Miller N. Essential Fatty Acid Plasma Profiles Following Gastric Bypass and Adjusted Gastric Banding Bariatric Surgeries. Obes Surg. 2016 Jun;26(6):1237-46. doi: 10.1007/s11695-015-1876-3. PMID 26328533